CLINICAL TRIAL: NCT06526585
Title: Examining the Immediate and Training Effects of Regular Stress Reduction Practices on Psychophysiological Markers of Anxiety
Brief Title: Stress Management Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Professor, Department of Psychiatry and Behavioral Sciences, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72131
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Stress; Anxiety
Keywords: Stress; Breathwork; Cyclic Sighing; Box Breathing; Hypnosis; Mood; Anxiety; Physiology; Heart Rate Variability; Respiratory Rate; fMRI; Brain Activity; Sleep
MeSH Terms: conditions — Anxiety Disorders | interventions — Hypnosis; Sound Recordings

STUDY DESIGN:
Intervention Model Description: Randomized prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cyclic Sighing Breathing (Experimental): Ten minutes a day of active breathwork practice for 28 days delivered remotely through a video link.
  Participants will also practice 10 minutes of active breathwork during the 2 MRI assessments, one before the start of the 28 days, and one after the completion of the 28 days.
  Interventions: Behavioral: Cyclic Sighing Breathing
- Box Breathing (Experimental): Ten minutes a day of active breathwork practice for 28 days delivered remotely through a video link.
  Participants will also practice 10 minutes of active breathwork during the 2 MRI assessments, one before the start of the 28 days, and one after the completion of the 28 days.
  Interventions: Behavioral: Box Breathing
- Hypnosis (Experimental): Ten minutes a day of hypnosis practice for 28 days delivered remotely through an audio link.
  Participants will also practice 10 minutes of hypnosis during the 2 MRI assessments, one before the start of the 28 days, and one after the completion of the 28 days
  Interventions: Behavioral: Hypnosis
- Audiobook on Stress (Active Comparator): Ten minutes a day of listening to sections of an audiobook about stress for 28 days (passive listening) delivered remotely through an audio link.
  Participants will also listen to the 10 minute segments during the 2 MRI assessments, one before the start of the 28 days, and one after the completion of the 28 days.
  Interventions: Behavioral: Audiobook

INTERVENTIONS:
Behavioral: Cyclic Sighing Breathing — Participants are instructed to be seated or lying down, and can keep their eyes open or closed throughout the 10 minutes of the breathing practice during the 28 days. Participants are instructed to keep their eyes closed when practicing the 10 minutes of the cyclic sighing during the 2 MRI assessments.
  The cyclic sighing protocol consists of a breathing pattern that involves inhaling deeply, starting abdominally, inhaling through the nose until lungs feel comfortably filled, immediately followed by a second shorter inhale, also through the nose, to maximally inflate the lungs. Then participants are instructed to slowly exhale through the mouth until their lungs feel empty. This cycle is repeated for 10 minutes.
  Arms: Cyclic Sighing Breathing
Behavioral: Box Breathing — Participants are instructed to be seated or lying down, and can keep their eyes open or closed throughout the 10 minutes of the breathing during the 28 days. Participants are instructed to keep their eyes closed when practicing the 10 minutes of the box breathing during the 2 MRI assessments.
  The CO2 tolerance test is done at baseline to determine their comfort level with the duration of each side of the box during box breathing.
  The box breathing protocol consists of a four-part breathing technique. The practice involves breathing through the nose in four equally timed parts: inhale, hold, exhale, and hold again, forming a 'box' of breaths (e.g. 4 sec inhale, 4 sec hold, 4 sec exhale, 4 sec hold).This cycle is repeated for 10 minutes.
  Arms: Box Breathing
Behavioral: Hypnosis — Participants are instructed to sit comfortably or lie down during the 28 day at home practice (Participants will be lying down in the scanner during the 2 MRIs). Then participants are asked to look up, slowly close their eyes, take a deep breath, slowly exhale, and let their body float, and then to imagine floating in a bath, a lake, a hot tub, or floating in space. Participants are then asked to picture an imaginary screen and visualize a place where it would naturally feel comfortable and relaxed. The participants then divide the screen in half and picture on the left side one thing that is causing them stress, with the rule that no matter what the participant picture, to keep their body comfortable and relaxed. Then on the right side of the screen the participants are asked to picture one thing that can be done about the problem on the left. At the end the participant will be guided to come out of the state of hypnosis. This exercise will take 10 minutes.
  Arms: Hypnosis
Behavioral: Audiobook — Participants are instructed to be seated or lying down, and can keep eyes open or closed throughout the 10 minutes of listening to the audiobook during the 28 days. Participants are instructed to keep their eyes closed during the 2 MRI assessments.
  Arms: Audiobook on Stress

SUMMARY:
This study will test the immediate and long term (post 4 weeks of daily practice) effectiveness of two breathwork practices, cyclic sighing and box breathing, in comparison to hypnosis and an audiobook about stress, on psychological and physiological variables.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* No contraindications to MRI imaging (like ferromagnetic metal in their body)

Exclusion Criteria:

* Pregnant or planning to get pregnant during study participation.
* Not able or willing to come to research location twice for MRI assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Neural Activation | Baseline Scan (Day 0) and and Follow-up Scan (From day 29 up to 4 weeks later, depending on the Scan scheduling availability)
  As measured for example by Fractional amplitude of low-frequency fluctuation (fALFF) signal, assessed using functional Magnetic Resonance Imaging (fMRI).

SECONDARY OUTCOMES:
Respiratory Rate | Daily from Baseline (Day 0) to a day prior to Endpoint (Day 28)
  Daily respiratory rate (RR) will be collected by WHOOP Strap 2.0, a wearable photoplethysmography (PPG) wrist sensor.
Heart Rate Variability | Immediate: Baseline Scan (Day 0) and Follow-up Scan (From day 29 up to 4 weeks later, depending on the Scan scheduling availability); Daily: from Baseline (Day 0) to a day prior to Endpoint (Day 28)
  Heart rate variability (HRV) will be measured in two modalities. Immediate continuous HRV, collected during resting-state MRI scans, will be measured by a wearable photoplethysmography (PPG) finger sensor. Daily HRV over the 28-day training period (RMSSD) will be collected by WHOOP Strap 2.0, a wearable PPG wrist sensor.
State Anxiety scale score | Immediate: Baseline Scan (Day 0) and Follow-up Scan (from day 29 up to 4 weeks later, depending on the Scan scheduling availability); Daily: from Baseline (Day 0) to a day prior to Endpoint (Day 28)
  The State-Trait Anxiety Inventory (STAI) is an instrument for measuring anxiety in adults. It has 2 scales: State Anxiety (S-Anxiety) and Trait Anxiety (T-Anxiety). The S-Anxiety scale measures anxiety due to temporary conditions, and the T-Anxiety measures anxiety on a general or more long-standing scale. The S-Anxiety is a 20-item scale; each item yields a score of 1 to 4. Scores on the STAI S-Anxiety scale increase in response to physical danger and psychological stress and decrease as a result of relaxation training.

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, MD, Principal Investigator — Stanford University
Locations (1):
- Psychiatry & Behavioral Sciences, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No